CLINICAL TRIAL: NCT02533089
Title: Training Lay Healthcare Workers to Optimize TB Care and Improve Outcomes in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dignitas International (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Lisa M Puchalski Ritchie, Dr., Unity Health Toronto
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: TB KT intervention
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KT intervention (Experimental): Multifaceted KT strategy employing peer-trainer led educational outreach, a point of care reminder tool, and a peer mentoring network.
  Interventions: Other: KT intervention
- Control (No Intervention): Control sites will receive no intervention, with LHW training left to the discretion of the health centers TB focus LHW. Control sites will not have access to the point of care tool.

INTERVENTIONS:
Other: KT intervention — Multifaceted KT intervention employing peer-trainer led educational outreach, a point of care reminder tool, and a peer mentoring network.
  Arms: KT intervention

SUMMARY:
Task shifting of less complex healthcare tasks to lay health workers (LHWs) is increasingly employed strategy to address the global shortage of skilled health workers. Despite availability of effective treatment, tuberculosis (TB) remains an important cause of mortality with 1.3 million lives lost globally to TB in 2012. The greatest proportion of new TB cases occurs in Africa and over 95% of TB deaths occur in low income countries (LICs). In response to the combined high TB burden and severe healthcare worker shortages in these settings, outpatient TB care is among the tasks commonly shifted to LHWs.

LHWs are community members who have received some training but are not healthcare professionals. Randomised trials show LHWs improve access to basic health services and TB treatment outcomes, however, insufficient training and supervision are recognized barriers to their effectiveness.

The investigators' goal is to improve TB care provided by LHWs in Malawi by implementing and evaluating a knowledge translation (KT) strategy designed to facilitate incorporation of evidence into LHW practice. The investigators will employ a mixed methods design including a pragmatic cluster randomized controlled trial to evaluate effectiveness of the strategy and qualitative methods to understand barriers and facilitators to scalability and sustainability of the program.

ELIGIBILITY:
Inclusion Criteria:

* all health centers in participating districts that routinely provide TB care will be included.
* LHWs who have received the intervention and patients receiving care at participating health centers will be eligible to participate in interviews

Exclusion Criteria:

* health centers that do not routinely provide TB care
* LHWs unwilling or unable to give informed consent.
* TB patients less than 18 years of age unaccompanied by a parent or guardian, patients/guardians or LHWs unwilling or unable to give informed consent, patients presenting to a health center they are not routinely followed at.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2016-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Puchalski Ritchie, MD,PhD, Principal Investigator — Li Ka Shing Knowledge Institute
Locations (1):
- 4 Districts, SE zone of Malawi (Balaka, Machinga, Mangochi, Mulanje), Malawi, Malawi, Malawi

REFERENCES:
- [Derived] Puchalski Ritchie LM, Kip EC, Mundeva H, van Lettow M, Makwakwa A, Straus SE, Hamid JS, Zwarenstein M, Schull MJ, Chan AK, Martiniuk A, van Schoor V. Process evaluation of an implementation strategy to support uptake of a tuberculosis treatment adherence intervention to improve TB care and outcomes in Malawi. BMJ Open. 2021 Jul 2;11(7):e048499. doi: 10.1136/bmjopen-2020-048499. PMID 34215610
- [Derived] Puchalski Ritchie LM, van Lettow M, Makwakwa A, Kip EC, Straus SE, Kawonga H, Hamid JS, Lebovic G, Thorpe KE, Zwarenstein M, Schull MJ, Chan AK, Martiniuk A, van Schoor V. Impact of a tuberculosis treatment adherence intervention versus usual care on treatment completion rates: results of a pragmatic cluster randomized controlled trial. Implement Sci. 2020 Dec 11;15(1):107. doi: 10.1186/s13012-020-01067-y. PMID 33308257
- [Derived] Puchalski Ritchie LM, van Lettow M, Makwakwa A, Chan AK, Hamid JS, Kawonga H, Martiniuk AL, Schull MJ, van Schoor V, Zwarenstein M, Barnsley J, Straus SE. The impact of a knowledge translation intervention employing educational outreach and a point-of-care reminder tool vs standard lay health worker training on tuberculosis treatment completion rates: study protocol for a cluster randomized controlled trial. Trials. 2016 Sep 7;17(1):439. doi: 10.1186/s13063-016-1563-2. PMID 27604571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 103 health centers enrolled, a total of 1153 patients
Pre-assignment Details: 109 health centers assessed for eligability, 6 health centers excluded as TB care not provided at the health center: all patients registered for TB care with treatment start and end dates within the study period included
Units Other Than Participants: health centers
Period: Overall Study
Arm/Group | KT Intervention | Control
Started | 605; 51 health centers | 548; 52 health centers
Completed | 364; 36 health centers (4 HC accrued no eligable patients 11 HC no patients with outcome data 241 cases missing outcome) | 434; 38 health centers (6 HC accrued no eligible patients 8 HC no patients with outcome data 114 cases missing outcome)
Not Completed | 241; 15 health centers | 114; 14 health centers

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KT Intervention | Control | Total
Number analyzed (Participants) | 605 | 548 | 1153
Age, Continuous [Mean (Full Range); unit: years] | 35.4 [0 to 94] | 36.3 [0 to 94] | 35.9 [0 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 273 | 227 | 500
  Male | 332 | 321 | 653
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
TB type = pulmonary TB [Count of Participants; unit: Participants] | 457 | 455 | 912

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Cases Successfully Treated, Defined as the Total Number of Cases Cured and Completing Treatment.
Description: primary outcome =proportion of cases successfully treated, defined as the total number of cases cured and completing treatment.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | KT Intervention | Control
Number analyzed (Participants) | 605 | 548
Participants | 297 | 348

2. Secondary Outcome: Proportion of Default Cases (Treatment Interrupted >= 2 Consecutive Months)
Description: secondary outcome =proportion of default cases (treatment interrupted >= 2 consecutive months)
Time Frame: 1 year
Population: analysis not conducted due to small proportion of default cases
Measure: Count of Participants; unit: Participants
Arm/Group | KT Intervention | Control
Number analyzed (Participants) | 605 | 548
Participants | 4 | 6

3. Secondary Outcome: Proportion of Successes Among HIV Co-infected Cases
Description: secondary outcome = proportion of successes among HIV co-infected cases
Time Frame: 1 year
Population: analysis not conducted due to large proportion of missing data
Measure: Count of Participants; unit: Participants
Arm/Group | KT Intervention | Control
Number analyzed (Participants) | 605 | 548
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Outcome data taken from ministry of health TB records, therefore only information of death during period of TB treatment available, no other adverse event data available
Arm/Group | KT Intervention | Control
All-Cause Mortality (participants affected / at risk) | 49/605 | 61/548
Serious Adverse Events (participants affected / at risk) | 0/605 | 0/548
Other Adverse Events (participants affected / at risk) | 0/605 | 0/548

LIMITATIONS AND CAVEATS:
outcome data limited to TB register outcome data.

give small number of defaults & high proportion of missing outcome data secondary outcomes not analyzed, factors related to missing outcome analyzed and included in primary analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT02533089/Prot_SAP_000.pdf